CLINICAL TRIAL: NCT00069940
Title: A Phase I Study Of Vaccination With Telomerase Peptide Plus GM-CSF
Brief Title: Vaccine Therapy and Sargramostim in Treating Patients With Sarcoma or Brain Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William Haining, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-365; P30CA006516 (NIH)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Brain and Central Nervous System Tumors; Gastrointestinal Stromal Tumor; Sarcoma
Keywords: adult glioblastoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; adult synovial sarcoma; childhood synovial sarcoma; childhood leiomyosarcoma; adult leiomyosarcoma; adult liposarcoma; childhood liposarcoma; gastrointestinal stromal tumor; recurrent childhood brain tumor; recurrent adult brain tumor; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; recurrent adult soft tissue sarcoma; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult oligodendroglioma; adult anaplastic oligodendroglioma; adult diffuse astrocytoma; adult mixed glioma; adult myxopapillary ependymoma; adult anaplastic ependymoma; childhood high-grade cerebral astrocytoma; recurrent childhood cerebral astrocytoma; untreated childhood cerebellar astrocytoma; recurrent childhood cerebellar astrocytoma; childhood infratentorial ependymoma; newly diagnosed childhood ependymoma; recurrent childhood ependymoma; childhood oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Gastrointestinal Stromal Tumors; Sarcoma; Glioblastoma; Sarcoma, Synovial; Leiomyosarcoma; Liposarcoma; Brain Neoplasms; Gliosarcoma; Astrocytoma; Oligodendroglioma; Glioma; Ependymoma; Familial ependymoma | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: sargramostim
Biological: telomerase: 540-548 peptide vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim increase the number of immune cells found in bone marrow or peripheral blood. Combining vaccine therapy with sargramostim may cause a stronger immune response and kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy when given together with sargramostim in treating patients with advanced sarcoma or brain tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of treatment with telomerase: 540-548 peptide vaccine and sargramostim (GM-CSF) in patients with sarcoma or brain tumor.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the frequency of T-cell specific vaccine antigens during and after administration of this regimen in these patients.
* Determine, preliminarily, the clinical response, if any, of patients treated with this regimen.

OUTLINE: Patients receive telomerase: 540-548 peptide vaccine subcutaneously (SC) on day 3 and sargramostim (GM-CSF) SC on days 1-4 of weeks 1, 3, 5, 7, 9, 11, 15, 19, and 23.

PROJECTED ACCRUAL: A total of 35 patients (20 adult and 15 pediatric) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following malignancies:

  * Stage III or IV sarcoma, including:

    * Leiomyosarcoma
    * Synovial cell sarcoma
    * Liposarcoma
    * Gastrointestinal stromal tumor
  * Brain tumor, including:

    * Diffuse pontine glioma*
    * Glioblastoma multiforme
    * Glialsarcoma NOTE: *For patients with diffuse pontine glioma, the requirement for histologic verification may be waived
* No known curative therapy
* HLA A*0201 positive by genotyping

PATIENT CHARACTERISTICS:

Age

* Over 2

Performance status

* Karnofsky 60-100% (patients over age 16)
* Lansky 60-100% (patients under age 16)

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* AST and ALT less than 2.5 times upper limit of normal (ULN)
* Bilirubin less than 1.5 times ULN

Renal

* Creatinine less than 1.5 times ULN

Cardiovascular

* No clinically significant cardiovascular disease

Pulmonary

* No clinically significant pulmonary disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior hematopoietic stem cell transplantation
* No other concurrent vaccine therapy
* No other concurrent immunotherapy

Chemotherapy

* No prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Concurrent dexamethasone allowed provided patient has been on a decreasing dose for the past 2 weeks and the current dose is the lowest clinically acceptable dose (ideally, less than 9-12 mg/day)

Radiotherapy

* No prior extensive-field radiotherapy that would compromise bone marrow function
* At least 2 weeks since prior local radiotherapy

Surgery

* At least 2 weeks since prior surgery

Other

* At least 2 weeks since prior imatinib mesylate
* No concurrent local anesthetic to administration site of vaccine

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2006-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Nicholas Haining, BM, BCh, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts, United States